CLINICAL TRIAL: NCT07369388
Title: Specular Endothelial Changes in Diabetic and Non-diabetic Patients Undergoing Phacoemulsification
Brief Title: Endothelial Changes in Diabetic and Non-diabetic Patients Undergoing Phacoemulsification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ehab Tharwat, Principal Invistigator, Al-Azhar University
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Endothelial Changes
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Endothelial Cell Density Loss
Keywords: Endothelial cell; Specular microscopy; Phacoemulsification
MeSH Terms: interventions — Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetic group (Active Comparator)
  Interventions: Procedure: Phacoemulsification
- Non-Diabetic group (Active Comparator)
  Interventions: Procedure: Phacoemulsification

INTERVENTIONS:
Procedure: Phacoemulsification — Cataract surgery using phacoemulsification is the most frequently performed ophthalmic procedure worldwide and is considered a highly effective and safe method for visual rehabilitation

SUMMARY:
The aim of this study is to evaluate and compare specular endothelial changes in diabetic and non-diabetic patients undergoing phacoemulsification by assessing endothelial cell density, coefficient of variation, and percentage of hexagonal cells preoperatively and postoperatively. This study also seeks to provide updated evidence on the influence of diabetes on corneal endothelial response to cataract surgery and to support evidence-based strategies for optimizing surgical outcomes

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years
* Presence of senile cataract suitable for phacoemulsification
* Clear cornea with no clinical signs of endothelial decompensation
* Ability to undergo specular microscopy examination
* For the diabetic group: confirmed diagnosis of type 2 diabetes mellitus

Exclusion Criteria:

* History of previous ocular surgery or trauma
* Corneal pathology affecting the endothelium
* Glaucoma or history of raised intraocular pressure
* Pseudoexfoliation syndrome
* Intraoperative complications

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-17 (Actual)

PRIMARY OUTCOMES:
Cell density | 1 week
Cell density | 1 month
Cell density | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar university, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided